CLINICAL TRIAL: NCT07294469
Title: Effect of Menthol on Motor Deficits and Sleep Disturbances in Patients With Parkinson's Disease
Brief Title: Menthol for Improving Movement and Sleep in Parkinson's Disease Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N202505079
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease
Keywords: Menthol; Parkinson's Disease; Motor Deficits; Sleep Disturbances
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol Group (Experimental): Participants in this arm will wear gloves and socks containing menthol daily for four weeks.
  Interventions: Drug: Menthol gloves and socks
- Placebo Group (Placebo Comparator): Participants in this arm will wear placebo gloves and socks daily for four weeks. These are identical in appearance and material to those used in the treatment group but contain no active menthol compound.
  Interventions: Drug: Placebo gloves and socks

INTERVENTIONS:
Drug: Menthol gloves and socks — Participants will wear menthol-containing gloves and socks for five minutes per day, five days a week, over a four-week period.
  Arms: Menthol Group
Drug: Placebo gloves and socks — Participants will wear gloves and socks with plain lotion for five minutes per day, five days a week, over a four-week period.
  Arms: Placebo Group

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disorder characterized by both motor and non-motor symptoms due to the degeneration of dopamine-producing neurons. There is currently no cure. Menthol, a natural compound that activates TRPM8 receptors, has shown neuroprotective and motor function benefits in preclinical PD models. In mice, distal limb immersion in menthol improved dopamine neuron survival and motor performance. Similar menthol-based interventions improved outcomes in a stroke model and a clinical trial with stroke patients. This study investigates whether topical menthol can offer therapeutic benefits for individuals with PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurological disorder that affects both motor and non-motor functions, with symptoms that can vary widely in severity. It is caused by the degeneration of dopamine-producing neurons in the substantia nigra, a brain region essential for movement control. The characteristic motor symptoms of PD include tremor, rigidity, bradykinesia, and postural instability. In addition to these motor impairments, many individuals with PD also experience non-motor symptoms, such as sleep disturbances, which can significantly impact their quality of life. Unfortunately, there is currently no cure for PD.

Menthol, a naturally occurring compound found in peppermint essential oil, has been shown to activate TRPM8 receptors in somatosensory neurons. Pharmacological activation of peripheral TRPM8 receptors enhances neural activity, which is subsequently transmitted to the brain.

In previous preclinical studies, the investigators used a dopamine toxin-induced PD mouse model and treated the mice with distal limb immersion in menthol. The results of immunohistochemical staining showed that limb immersion in menthol reduced the loss of dopamine neurons and increased the dopamine content in the mouse striatum. The mice's motor function also improved, as indicated by a significant increase in the time they spent running on the rotarod. The investigators also evaluated the effects of menthol in a stroke mouse model induced by MCAO. Topical application of menthol to the paw alleviated acute cerebral infarction and ischemia-induced sensorimotor deficits in MCAO mice.

In our recent clinical trial, the investigators evaluated the effects of menthol-containing gloves and socks in acute ischemic stroke patients. After four weeks of treatment, patients showed improvements in their Modified Rankin Scale (mRS) and Barthel Index (BI) scores, suggesting that this intervention may help enhance functional recovery. Based on these promising results, the investigators hypothesize that a similar approach could benefit individuals with PD.

The investigators aim to conduct a double-blind, randomized controlled trial evaluating the effectiveness of menthol-containing gloves and socks in treating motor deficits and sleep disorders in patients with PD：A total of 80 patients with PD will be randomized into the following groups: (1) menthol-containing gloves and socks (2) placebo. The treatment duration will be 4 weeks, with 4 weeks follow-up. All patients will be clinically assessed at the randomization, 4 and 8 week. Unified Parkinson's Disease Rating Scale (UPDRS) I,II,III, Pittsburgh Sleep Quality Index (PSQI), Parkinson's Disease Sleep Scale-2 (PDSS-2), Parkinson's Disease Questionnaire (PDQ-39) and detailed neurological examination will be included in the assessment.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 30 and 80 years (inclusive);
2. diagnosed with idiopathic PD based on the Brain Bank criteria of the UK Parkinson's Disease Society less than 3 years;
3. Hoehn and Yahr stages 1-3 and currently receiving treatment; experiencing sleep disorders with a Pittsburgh Sleep Quality Index (PSQI) > 5;
4. has signed the informed consent form approved by the Institutional Review Board and dated accordingly;
5. no changes in PD medications within four weeks prior to participating in this trial, and no dosage changes during the study period;
6. able to use other medications that may affect sleep, except those explicitly prohibited, provided the dosage has been stable for the four weeks before screening and remains unchanged during the study.

Exclusion Criteria:

1. menthol allergy;
2. pregnant and breastfeeding women;
3. diagnosed with secondary and atypical PD;
4. patients with conditions such as uremia, cirrhosis, congestive heart failure with pulmonary edema, coagulation disorders, epilepsy, alcoholism, drug abuse, or
5. deemed unsuitable for participation in this study by the principal investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) I,II,III | Evaluations will be conducted at the time of randomization and will serve as baseline data.
  The UPDRS is a clinical tool to assess the severity of Parkinson's disease. It consists of:
  Part I: Mentation, Behavior, and Mood (cognitive and psychiatric symptoms); Part II: Activities of Daily Living (self-reported motor activities); Part III: Motor Examination (clinician-assessed motor symptoms); The combined score of Parts I, II, and III reflects overall disease severity.
Unified Parkinson's Disease Rating Scale (UPDRS) I,II,III | Evaluations will be conducted at the fourth week after the start of the intervention.
  The UPDRS is a clinical tool to assess the severity of Parkinson's disease. It consists of:
  Part I: Mentation, Behavior, and Mood (cognitive and psychiatric symptoms); Part II: Activities of Daily Living (self-reported motor activities); Part III: Motor Examination (clinician-assessed motor symptoms); The combined score of Parts I, II, and III reflects overall disease severity.
Unified Parkinson's Disease Rating Scale (UPDRS) I,II,III | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention.
  The UPDRS is a clinical tool to assess the severity of Parkinson's disease. It consists of:
  Part I: Mentation, Behavior, and Mood (cognitive and psychiatric symptoms); Part II: Activities of Daily Living (self-reported motor activities); Part III: Motor Examination (clinician-assessed motor symptoms); The combined score of Parts I, II, and III reflects overall disease severity.
Pittsburgh Sleep Quality Index (PSQI) | Evaluations will be conducted at the time of randomization and will serve as baseline data.
  The PSQI is a self-report questionnaire assessing sleep quality and disturbances over the past month. It consists of 19 items across 7 domains: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
Pittsburgh Sleep Quality Index (PSQI) | Evaluations will be conducted at the fourth week after the start of the intervention.
  The PSQI is a self-report questionnaire assessing sleep quality and disturbances over the past month. It consists of 19 items across 7 domains: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
Pittsburgh Sleep Quality Index (PSQI) | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention.
  The PSQI is a self-report questionnaire assessing sleep quality and disturbances over the past month. It consists of 19 items across 7 domains: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.

SECONDARY OUTCOMES:
Parkinson's Disease Sleep Scale-2 (PDSS-2) | Evaluations will be conducted at the time of randomization and will serve as baseline data.
  The PDSS-2 is a self-reported tool designed to assess sleep disturbances specifically in individuals with Parkinson's disease. It includes 15 items covering various sleep-related issues such as sleep onset, duration, nocturnal motor symptoms, and daytime sleepiness.
Parkinson's Disease Sleep Scale-2 (PDSS-2) | Evaluations will be conducted at the fourth week after the start of the intervention.
  The PDSS-2 is a self-reported tool designed to assess sleep disturbances specifically in individuals with Parkinson's disease. It includes 15 items covering various sleep-related issues such as sleep onset, duration, nocturnal motor symptoms, and daytime sleepiness.
Parkinson's Disease Sleep Scale-2 (PDSS-2) | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention.
  The PDSS-2 is a self-reported tool designed to assess sleep disturbances specifically in individuals with Parkinson's disease. It includes 15 items covering various sleep-related issues such as sleep onset, duration, nocturnal motor symptoms, and daytime sleepiness.
Parkinson's Disease Questionnaire (PDQ-39) | Evaluations will be conducted at the time of randomization and will serve as baseline data.
  The PDQ-39 is a 39-item self-report questionnaire designed to assess health-related quality of life in people with Parkinson's disease. It covers 8 domains: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and sleep.
Parkinson's Disease Questionnaire (PDQ-39) | Evaluations will be conducted at the fourth week after the start of the intervention.
  The PDQ-39 is a 39-item self-report questionnaire designed to assess health-related quality of life in people with Parkinson's disease. It covers 8 domains: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and sleep.
Parkinson's Disease Questionnaire (PDQ-39) | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention.
  The PDQ-39 is a 39-item self-report questionnaire designed to assess health-related quality of life in people with Parkinson's disease. It covers 8 domains: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hung Chen, PhD, Study Director — International Master Program in Integrative Health, College of Chinese Medicine, China Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data including paper and electronic files will be destroyed after two years since the end of the study. Data obtained from the study, if digitized, will be stored on the investigator's computer in the hospital office and secured the password. Written data will be kept in a locked drawer in the investigator's office and stored separately from the subject's consent form. The data will be kept for five years after the end of the trial, at which time the digital data will be deleted from the computer and the written data will be deleted by shredder.

REFERENCES:
- [Background] Huang SS, Su HH, Chien SY, Chung HY, Luo ST, Chu YT, Wang YH, MacDonald IJ, Lee HH, Chen YH. Activation of peripheral TRPM8 mitigates ischemic stroke by topically applied menthol. J Neuroinflammation. 2022 Jul 27;19(1):192. doi: 10.1186/s12974-022-02553-4. PMID 35897101